CLINICAL TRIAL: NCT00211315
Title: Treatment of Congenital Telangiectasia (Coat's Disease) With Open-label Anecortave Acetate (15mg.)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Alcon Research (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA in Coat's Disease
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Coat's Disease
MeSH Terms: conditions — Retinal Telangiectasis | interventions — anecortave acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: anecortave acetate

SUMMARY:
Congenital Telangiectasia or Coat's disease is an uncommon disorder that involves the growth of blood vessels of the macula. These blood vessels msy extend beneth the retina to produce an area of sub-retinal neovascularization(growth of abnormal blood vessels under the retina which "leak" fluid, causing reduction in vision). Limited forms of treatment are available in managing the neovascularization and its consequences. Anecortave Acetate injection will be considered as an attempt to control the growth of the abnormal blood vessels.

DETAILED DESCRIPTION:
After evaluation, the patient will receive an injection of anecortave acetate (15mg) juxtascleral with a special cannula in the study eye. the patient will be contacted via phone on the day following the injection. If problem arises patient has to come back to see the study doctor. if patient is stable, a 3 month follow-up visit will be st-up.if the patient does not show improvement, the patient may be offered either thermal laser or PDT. If patient is stable, on the month 6 visit ,the patient will again receive another injection of anecortave acetate. The succeding follow-up schedule will be followed for a total of 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of congenital Telangiectasia (Coat's Disease).
2. Patients must be 18 years of age or older to receive treatment.
3. Visual acuity of 20/30 to 20/320 Study Eye on the ETDRS visual acuity chart.
4. Visual acuity of 20/800 or better Fellow Eye on the ETDRS visual acuity chart.

Exclusion Criteria:

1. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
2. Patients who have undergone intraocular surgery within last 2 months.
3. Patient participating in any other investigational drug study.
4. Use of an investigational drug or treatment related or unrelated to their condition within 30 days prior to receipt of study medication.
5. Inability to obtain photographs to document CNV (including difficulty with venous access).
6. Patient with significant liver disease or uremia.
7. Patient with known adverse reaction to fluorescein and indocyanine green or iodine.
8. Patient has a history of any medical condition which would preclude scheduled visits or completion of study.
9. Patient has had insertion of scleral buckle in the study eye
10. Patient has received radiation treatment.
11. Patient is on anticoagulant therapy with the exception of aspirin.
12. Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2002-03; Study Completion 2007-03

PRIMARY OUTCOMES:
to investigate the use of anecortave acetate in coats's disease | 24 months

SECONDARY OUTCOMES:
mean change in ETDRS visual acuity , OCT, leakage in FA compared at baseline at month 24. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A. Yannuzzi, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States